CLINICAL TRIAL: NCT03329911
Title: A Multicenter, Randomized, Double Blind, Phase III Study of BAT1706 Versus EU Avastin® Plus Chemotherapy in Patients With Advanced Non Squamous Non Small Cell Lung Cancer
Brief Title: A Comparative Study of BAT1706 and EU Avastin® in Patients With Advanced Non Squamous Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAT1706-003-CR
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EU Avastin® (Active Comparator): Drug:EU Avastin® 15 mg/kg IV infusions ,every 3 weeks of a cycle for up to 6 cycles, followed for those with non-progressive disease with maintenance monotherapy with Bevacizumab-EU up to a maximum of 8 months.
  Drug: Paclitaxel 200mg/m² via IV infusions, every 3 weeks of a cycle for up to 6 cycles
  Drug: Carboplatin AUC 6.0 mg/mL•minute via IV infusions,every 3 weeks of a cycle for up to 6 cycles
  Interventions: Drug: EU Avastin®; Drug: Paclitaxel; Drug: carboplatin
- BAT1706 (Experimental): BAT1706 15 mg/kg IV infusions ,every 3 weeks of a cycle for up to 6 cycles, followed for those with non-progressive disease with maintenance monotherapy with BAT1706 up to a maximum of 8 months.
  Drug: Paclitaxel 200mg/m² via IV infusions, every 3 weeks of a cycle for up to 6 cycles
  Drug: Carboplatin AUC 6.0 mg/mL•minute via IV infusions,every 3 weeks of a cycle for up to 6 cycles
  Interventions: Drug: BAT1706; Drug: Paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: EU Avastin® — 100 mg/4 mL
  Arms: EU Avastin®
Drug: BAT1706 — 100 mg/4 mL
  Arms: BAT1706
Drug: Paclitaxel — 200 mg/m²
Drug: carboplatin — target area under the curve [AUC] 6 mg/mL•minute

SUMMARY:
This is a Phase III, randomized, double blind, multicenter, active comparator, parallel two arm study to compare the efficacy, and to evaluate the safety, and immunogenicity of BAT1706 to EU Avastin® in patients with previously untreated advanced non-squamous non-small cell lung cancer (nsNSCLC) to demonstrate clinical equivalence of BAT1706 and EU Avastin®.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV nsNSCLC or recurrent disease (any Stage at initial diagnosis) no longer amenable to curative surgery or local therapy (histologically or cytologically confirmed).
2. No prior systemic therapy for metastatic disease. Prior systemic therapy and/or radiotherapy for locally advanced disease is permitted if completed ≥ 6 months prior to randomization.
3. Tumors without activating EGFR or ALK mutation. Patients with unknown mutation status or known activating EGFR or ALK mutation may be included provided the corresponding targeted agent is not available and chemotherapy is the standard of care of the study center.
4. At least one measurable target lesion according to RECIST 1.1 (Appendix 13.4) as confirmed by CIR; bone only and brain-only metastases are not allowed. Lesions previously treated with radiotherapy are non-target lesion.
5. Eastern Cooperative Oncology Group performance status of 0 or 1 and life expectancy > 3 months based on Investigator's judgment.

Exclusion Criteria:

1. Diagnosis of small cell carcinoma of the lung, mixed predominant squamous cell carcinoma of the lung, NSCLC not otherwise specified.
2. Tumor cavitation, tumor invading into large blood vessels or close to large vessels with an increased risk of bleeding, according to Investigator's judgment.
3. Prior therapy with monoclonal antibodies or small molecule inhibitors against VEGF or VEGFR, including Avastin®.
4. Prior systemic therapy for metastatic disease.
5. Prior systemic anticancer therapy, or radiotherapy for locally advanced nsNSCLC if completed < 6 months prior to screening.
6. Previous malignancy other than NSCLC in the last 5 years except for basal cell cancer of the skin or pre invasive cancer of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shengfeng Li, Study Director — Sponsor GmbH
Locations (5):
- The First Affiliated Hospital of Xiamen University, Xiamen, China
- Clinical Medical Research S.C., Orizaba, Mexico
- National Hospital Oncology, Bloemfontein, South Africa
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)
- CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- EU Avastin®: Drug:EU Avastin® 15 mg/kg IV infusions ,every 3 weeks of a cycle for up to 6 cycles, followed for those with non-progressive disease with maintenance monotherapy with Bevacizumab-EU up to a maximum of 8 months.
  Drug: Paclitaxel 200mg/m² via IV infusions, every 3 weeks of a cycle for up to 6 cycles
  Drug: Carboplatin AUC 6.0 mg/mL•minute via IV infusions,every 3 weeks of a cycle for up to 6 cycles
  EU Avastin®: 100 mg/4 mL
  Paclitaxel: 200 mg/m²
  carboplatin: target area under the curve [AUC] 6 mg/mL•minute
- BAT1706: BAT1706 15 mg/kg IV infusions ,every 3 weeks of a cycle for up to 6 cycles, followed for those with non-progressive disease with maintenance monotherapy with BAT1706 up to a maximum of 8 months.
  Drug: Paclitaxel 200mg/m² via IV infusions, every 3 weeks of a cycle for up to 6 cycles
  Drug: Carboplatin AUC 6.0 mg/mL•minute via IV infusions,every 3 weeks of a cycle for up to 6 cycles
  BAT1706: 100 mg/4 mL
  Paclitaxel: 200 mg/m²
  carboplatin: target area under the curve [AUC] 6 mg/mL•minute
Period: Overall Study
Arm/Group | EU Avastin® | BAT1706
Started | 326 | 325
Completed | 209 | 222
Not Completed | 117 | 103

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EU Avastin® | BAT1706 | Total
Number analyzed (Participants) | 326 | 325 | 651
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 208 | 233 | 441
  >=65 years | 118 | 92 | 210
Age, Continuous [Median (Full Range); unit: years] | 60 [26 to 88] | 61 [27 to 84] | 61 [26 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 97 | 194
  Male | 229 | 228 | 457
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 11 | 24
  Asian | 140 | 141 | 281
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 171 | 172 | 343
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 67 | 64 | 131
  China | 139 | 140 | 279
  Ukraine | 98 | 102 | 200
  South Africa | 6 | 2 | 8
  Mexico | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary efficacy endpoint is ORR at Week 18 (ORR18) based on tumor response evaluated according to RECIST 1.1 as assessed by CIR. Each patient will be assigned to one of the following RECIST 1.1 categories based on independent CIR, irrespective of protocol deviations or missing data:
  CR: complete response. PR: partial response. SD: stable disease. PD: progressive disease. NE: not evaluable (insufficient data)
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | EU Avastin® | BAT1706
Number analyzed (Participants) | 326 | 325
Participants | 156 | 145

2. Secondary Outcome: Progression Free Survival Rate
Description: Progression free survival rate at 12 months, defined as the proportion of patients being alive without documented progression 12 months after randomization, using Kaplan-Meier method.
Time Frame: 8 months,1 year and 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Progression Free Survival Time
Description: Progression free survival time defined as the time from the date of randomization to the date of documented clinical or radiological progression or death due to any cause using Kaplan-Meier method.
Time Frame: 8 months,1 year and 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate at 12 months, defined as the proportion of patients being alive 12 months after randomization using Kaplan-Meier method.
Time Frame: 8 months,1 year and 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival Time
Description: Overall survival time defined as the time from randomization to death of any cause using Kaplan-Meier method.
Time Frame: 8 months,1 year and 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Response Rate
Description: ORR at Week 6 (ORR6) and ORR at Week 12 (ORR12), based on tumor response as assessed by CIR, and best ORR of confirmed responses at end of study assessed by local radiologist/Investigator if after Week 18 according to RECIST 1.1.
Time Frame: Week 6 and Week 12
Reporting Status: Not Posted

7. Secondary Outcome: Duration of Response
Description: Duration of response defined as the time from first documentation of a response (CR or PR) and the first documentation of progression (assessed by local radiologist/Investigator if after Week 18) according to RECIST 1.1.
Time Frame: 8 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Plasma Level of Anti Drug Antibodies (ADA) and Neutralizing Anti-drug Antibodies (NADA) Correlated With Bevacizumab Plasma Level
Description: Plasma level of anti drug antibodies (ADA) and neutralizing anti-drug antibodies (NADA) correlated with bevacizumab plasma level
Time Frame: 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Bevacizumab Plasma Exposure Following Treatments of BAT1706 or EU Avastin®
Description: Bevacizumab plasma exposure following treatments of BAT1706 or EU Avastin®
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of the first study medication administration until 28 days after discontinuation/completion of the study medication or up to Week 53 after randomization- All AEs, regardless of relationship to the study medication/study procedures. During the LTE study, only adverse events of special interest (AESIs) and SAEs until 28 days after the subject's last dose will be collected.
Arm/Group | EU Avastin® | BAT1706
All-Cause Mortality (participants affected / at risk) | 4/324 | 7/325
Serious Adverse Events (participants affected / at risk) | 119/324 | 119/325
Other Adverse Events (participants affected / at risk) | 8/324 | 9/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EU Avastin® (N=324) | BAT1706 (N=325)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 46 | 31
Infections and infestations (Infections and infestations) | 22 | 27
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 19 | 21
Gastrointestinal disorders (General disorders) | 12 | 12
Cardiac disorders (Cardiac disorders) | 4 | 11
Vascular disorders (Vascular disorders) | 8 | 5
General disorders and administration site conditions (Gastrointestinal disorders) | 4 | 8
Nervous system disorders (Nervous system disorders) | 4 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EU Avastin® (N=324) | BAT1706 (N=325)
Neoplasms benign, malignant and unspecified (inclcysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hepatobiliarydisorders (Hepatobiliary disorders) | 1 | 1
Renal and urinary disorders (Renal and urinary disorders) | 2 | 3
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03329911/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03329911/SAP_003.pdf